CLINICAL TRIAL: NCT00422370
Title: Lipid Based Food Additives for Treating Patients With Dry Mouth
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hadassah Medical Organization (Other)
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: 38-29.12.06
Record Dates: First submitted 2006-12-14; First posted 2007-01-17 (Estimated); Last update posted 2007-01-17 (Estimated); Status verified 2006-12

CONDITIONS: Xerostomia
MeSH Terms: conditions — Xerostomia

INTERVENTIONS:
Device: lipid based additives based on vegetable oil & lecithin

SUMMARY:
Over 10% of adult population suffers from dry mouth (xerostomia). The aim of this double blind prospective clinical trial is to examine a new lipid based food additive formulation to ease mouth dryness in these patients.

ELIGIBILITY:
Inclusion Criteria:

* Dry mouth patients

Exclusion Criteria:

* Disabled patients
* Pregnant
* Full upper denture
* Under 18 years old

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2007-01

PRIMARY OUTCOMES:
Improvement in dry mouth symptom

CONTACTS AND LOCATIONS:
Overall Officials: Doron J Aframian, DMD PhD, Study Chair — Reference: Kelly HM et al. Bioadhesive,rheological, lubricant and other aspectes of an oral gel formulation intended for the treatment of xerostomia. Int J Phramac. 2004; 278: 391-406; Doron J Aframian, DMD PhD, Study Chair — Salivary Gland Clinic, Department of Oral Medicine The Hebrew University-Hadassah School of Dental Medicine Jerusalem, Israel P.O.B 12272, Zip code 91120